CLINICAL TRIAL: NCT05080322
Title: A Randomized, Open-labeled, Multicenter Clinical Trial to Compare the Efficacy and Safety of On-demand and Continuous Administration of Nasal Spray in the Treatment of Moderate-to-severe Persistent Allergic Rhinitis
Brief Title: Efficacy and Safety of On-demand and Continuous Administration of Nasal Spray in the Treatment of Allergic Rhinitis
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Zheng Liu ENT (Other)
Collaborators: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Zhongnan Hospital (Other); The People's Hospital of Hebei Province (Other)
Responsible Party: Sponsor-Investigator, Zheng Liu ENT, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: AR-DEM-2021
Record Dates: First submitted 2021-07-27; First posted 2021-10-15 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Fluticasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- on-demand intranasal corticosteroid (INS) plus antihistamines (AH1) (Experimental): the patients will be treated with on-demand intra-nasal corticosteroid (INS) plus antihistamines (AH1) for 4 weeks
  Interventions: Drug: Fluticasone Nasal 50 Mcg/Inh Nasal Spray, Azelastine Nasal 140 Mcg/Inh Nasal Spray
- on-demand intranasal corticosteroid (INS) (Experimental): the patients will be treated with on-demand intra-nasal corticosteroid (INS) for 4 weeks
  Interventions: Drug: Fluticasone Nasal 50 Mcg/Inh Nasal Spray
- maintenance intranasal corticosteroid (INS) (Active Comparator): the patients will be treated with intra-nasal corticosteroid(INS) maintenance therapy for 4 weeks
  Interventions: Drug: Fluticasone Nasal 50 Mcg/Inh Nasal Spray

INTERVENTIONS:
Drug: Fluticasone Nasal 50 Mcg/Inh Nasal Spray, Azelastine Nasal 140 Mcg/Inh Nasal Spray — on-demand INS (Fluticasone) combined with nasal spray AH1(Azelastine)
  Other Names: Flixonase,H20140117, AZEP,H20150201
  Arms: on-demand intranasal corticosteroid (INS) plus antihistamines (AH1)
Drug: Fluticasone Nasal 50 Mcg/Inh Nasal Spray — on-demand or maintenance
  Other Names: Flixonase,H20140117
  Arms: maintenance intranasal corticosteroid (INS); on-demand intranasal corticosteroid (INS)

SUMMARY:
WHO recommend to divide AR into 4 subgroups according to the symptom frequency (intermittent or persistent) and severity (mild or moderate-to-severe). For the persistent moderate-to-severe AR subgroup, the guideline suggests to treat with intranasal corticosteroid (INS) plus antihistamines (AH1) for 2-4 weeks. If the symptom is controlled then degrade the treatment (usually with INS) and maintenance for more than 4 weeks. However, up to 70% of patients suffering from AR do not follow treatment recommendation, they stopped medication when they feel better. This behavior always leads to uncontrolled AR, which has been identified as a high-risk factor of induction and exacerbation of asthma and chronic rhinosinusitis. A recent survey showed that AR patients prefer to an on-demand treatment rather than continuous treatment. In general, poor adherence is always a considerable issue for all long-term treatments. Previous studies have shown that as dosing frequency increases, the adherence rate decreases. Thus, less medication frequency is an important factor to optimize the management of chronic diseases including AR.

Intranasal AH1 can relieve AR symptoms including sneezing, rhinorrhea and nasal itching in 3 to 5 minutes, while INS can inhibit the underlying mucous allergic inflammation and is recommended as the first-line medication for moderate-to-severe AR. INS combined AH1 have shown a synergic effect on control AR inflammation and provide rapid AR symptom relief. Investigators hypothesis that the on-demand administration of INS combined AH1 can achieve similar AR control level with less dosing frequency as compared to the daily INS maintenance in controlled moderate-to-severe AR patients.

DETAILED DESCRIPTION:
Background/Significance The prevalence of AR is increasing worldwide. A large number of studies have shown that AR has a significant adverse impact on the quality of life especially in the moderate-to-severe AR population. However, as AR is not a fatal disease, only a small proportion of AR patients will go to hospital to seek professional medical advice. They have a tendency to do so only when their AR-related symptoms become intolerable, which led to a dramatic low level of AR control. It is well known that uncontrolled AR has been identified as a high-risk factor of exacerbation of asthma and chronic rhinosinusitis. In AR patients, 40% will develop asthma and up to 30% will develop chronic sinusitis. Adequate treatment of AR always help to improve patients' quality of life and also reduce the risk of AR related complications.

To achieve the goal of AR control, long-term treatment is always needed. AR is an IgE-mediated inflammatory disease induced by allergen exposure. Our previous study had shown that more than 90% of AR patients in central China were induced by house dust mite (HDM), a perennial indoor allergen. HDM exposure leads to persistent allergic inflammation in nasal mucous and causes periodic exacerbation of AR symptoms. INS is currently the cornerstone medication to inhibit the allergic inflammation and is recommended as the first-line medication for moderate-to-severe AR. However, the anti-inflammation effect can only be achieved after administrate for several days to two weeks. For this reason, the ARIA guideline suggests to use INS regularly for 2-4 weeks, then step down gradually. In another side, antihistamine belongs to symptom-relief medication, which has been proven to act within 5min for nasal spray and 30min for oral route. Antihistamine is also recommended as first-line medication for mild AR patients and combined with INS for moderate-to-severe AR patients. Our previous studies had shown that if AR patients were treated according to the current guideline for 15 days, only 72.3% of them were controlled. However, if the treatment extended to 60 days, more than 95% would achieve AR controlled.

Low adherence is always a considerable issue for long-term treatment. In asthma patients, more than 80% of patients taken β2 agonist as needed to relieve their symptom instead of daily using inhalant corticosteroids. For AR, the adherence to treatment recommendation was below 30% in the real world. Most AR patients wouldn't take their medication continuously for 14 days as they usually suffered from several episodes of short-term AR symptoms. They have a strong preference for a treatment which can provide both a rapid onset of action and clinically-relevant symptom relief.

In this study, investigators will compare the AR control level of on-demand treatment versus daily maintenance treatment in moderate-to-severe AR patients. If the on-demand treatment can achieve similar or non-inferior AR control rate as daily maintenance treatment, it will be very helpful to optimize current management of AR patients.

Preliminary Data A recent study in 150 pollen-induced AR children found that the percentage of symptom-free-day was in favor of INS on-demand (30%) compared with low dosage INS daily (22%), although the statistical significance was not achieved. It implied that on-demand fluticasone propionate treatment was at least as effective as a regular treatment at a lower dose. The authors concluded that an on-demand INS strategy has the advantage of a lower overall corticosteroid exposure and less costs.

Two large randomized controlled studies in mild asthma patients (4215 and 3849 patients were randomized respectively) also shown that budesonide-formoterol used as needed was non-inferior to twice-daily budesonide with respect to the rate of severe asthma exacerbations during 52 weeks of treatment.

Investigators have validated the Allergic Rhinitis Control Test (ARCT) questionnaire in 255 AR Chinese patients, the ARCT score ≥20 was regard as controlled AR. Investigators also validated ARCT questionnaire in guiding stepwise treatment in 510 AR patients. Thus, the ARCT questionnaire will be used to calculate the AR control level in our study. In our randomized controlled trial, 129 AR patients received INS without dosage adjustment for 60 days, 85.8% were controlled AR (ARCT score≥20). In a hospital based study, investigators found that only 4.8% of the AR patients were controlled without taken medication or taken medication occasionally. However, the data could not reflect the real-life situation as usually only the intolerable symptoms would drive AR patients to the hospital. There is still lack of data of AR control rate in on-demand treatment patients.

Research Design and Methodology Study Design This is an open-labeled, randomized, controlled clinical study with HDM-related AR which will be conducted in four multicenter in Central China.. The symptom uncontrolled moderate-severe AR patient were enrolled with ARCT˂20. In the run-in period, AR patients will be treated with INS plus AH1 twice daily for 2 weeks and assessed with ARCT questionnaire and Quality-of-Life Questionnaires. If AR is controlled, the patients will be randomized into on-demand INS combine intranasal AH1 group, on-demand INS or daily INS maintenance group and treat for 4 weeks, then the treatment will be stopped and the patients will be followed up for another 8 weeks. During the study period, the patients have to fill in the diary card every day to record TNSS and daily ARCT every day. During the run-in period, the treatment and follow-up period, the patients were followed up every 4 weeks in the hospital to finish ARCT, RQLQ and IPQ questionnaires to compare the AR control and recurrence time among the three groups.

Study Population This is a multi-center study. Patients with persistent moderate-to-severe AR will be enrolled after sign the informed and content form, adolescents need guardian consent.

Inclusion Criteria (1) 18-65 years old（2) AR patients (according to ARIA guidelines)（3) Mono-sensitized to HDM and had AR symptoms after HDM exposure; （4) had at least 2 nasal symptoms(sneezing, runny nose, itching, nasal congestion) in the screening period（4) ARCT score ≥20 after 2-week INS combined with AH1 treatment at run-in period（5) had adequent informed and given their consent to participate in the study.

Exclusion Criteria

(1) Pregnant or lactating women, patients with malignant tumor, patients with congenital or acquired immunodeficiency disease, patients with mental illness（2) Acute upper respiratory infection in the run-in period（3) History of chronic sinusitis with nasal polyps（4) Severe deviation of nasal septum（5) received allergen immunotherapy in the past 5 years（6) received biological therapy in the past 6 months （7)Acute upper respiratory tract infection in run-in period（8) Patients who failed to achieve AR control in the run-in period.(9) Patients who are participating in other clinical trials; (10) patients who are not suitable for this clinical trial due to other reasons (evaluated by investigators).

Study protocol

1. Enroll HDM mono-sensitized AR patients.
2. Diagnosis and differential diagnosis were made according to ARIA. The other related diseases that may increase nasal symptoms were excluded according to ARIA.
3. Evaluate ARCT score, RQLQ, and Brief IPQ questionnaire in the baseline. Treat with intranasal Azelastine and Fluticasone Propionate and re-evaluate ARCT score to assure ARCT≥20 after 2 weeks, before randomization. During the run-in period the patients need to complete the daily TNSS and the daily ARCT on-line.
4. Randomize into On-demand intranasal Azelastine and Fluticasone Propionate group, on-demand Fluticasone Propionate group or daily intranasal Fluticasone maintenance group. The patients have to complete the dairy online to record the TNSS and ARCT.
5. The pharmacotherapy will be stopped after 4 weeks and the patients will be followed up for another 8 weeks. During the follow-up period, the patients filled the diary card every day to recorded TNSS and ARCT. During the treatment and follow-up period, the patients have to revisit every 4 weeks in the hospital. ARCT, RQLQ and IPQ questionnaires were filled in to compare the AR control and recurrence time among the three groups.

Statistical Approach and sample size calculation Referring to the relevant literature, investigators assume the AR control rate of continuous NCS treatment group will be 85% and the AR control rates of on-demand NCS group and on-demand NCS + AH1 group both will be 75%, investigators also set the non-inferiority margin value as 10%, and the enrollment ratio as 1:1:1. The sample size of each group is 49, plus 20% drop-out rate, a total of 180 cases are required in this trial.

Possible risks and preventive measures Fluticasone propionate nasal spray and azelastine hydrochloride nasal spray used in this study have been approved and widely used in AR patients for many years in China. The common local adverse reactions include epistaxis, nasal cavity and throat dryness, local nasal pain and irritation, bitter taste or nausea, etc. Systemic adverse reactions are rare. Any adverse events will be recorded and managed by the investigators according to Good Clinical Practice guidelines.

Data collection and statistical analysis Data collection: the patients filled in the diary on-line every day to record the nasal symptom (TNSS) score and ARCT. The symptoms included nasal itching, sneezing, runny nose and nasal congestion. The scoring criteria were: 0: asymptomatic, 1: mild, 2: moderate and 3: severe. The ARCT score was used to assess the control of AR symptoms. During the treatment and follow-up period, the patients were followed up every 4 weeks on-site. ARCT, RQLQ and IPQ questionnaires were filled in to compare the AR control and recurrence among the three groups.

Statistical analysis: the primary endpoint was AR control level at 4-week among the treatment groups. The secondary endpoint included TNSS scores of different treatment groups, AR recurrence time after treatment, RQLQ and IPQ questionnaire score comparison and adverse events among different treatment groups. The data of continuous variables were tested for normality, and the variables in accordance with normal distribution were expressed by mean ± standard deviation. T test was used to compare the differences between groups; The variables of non-normal distribution were expressed by median ± quartile interval. Mann Whitney U test was used to compare the differences between groups; For binary variables, Chi square test was used to determine the difference between groups. Kaplan Meier survival curve was used to analyze the recurrence time of AR in different treatment groups. A p value less than 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* AR patients (according to ARIA guidelines)
* Mono-sensitized to HDM and had AR symptoms after HDM exposure;
* Participants had at least 2 nasal symptoms(sneezing, runny nose, itching, nasal congestion) in the screening period
* ARCT score ≥20 after 2-week INS combined with AH1 treatment at run-in period
* had adequent informed and given their consent to participate in the study.

Exclusion Criteria:

* Pregnant or lactating women, patients with malignant tumor, patients with congenital or acquired immunodeficiency disease, patients with mental illness
* Acute upper respiratory infection in the run-in period
* History of chronic sinusitis with nasal polyps
* Severe deviation of nasal septum
* received allergen immunotherapy in the past 5 years
* received biological therapy in the past 6 months
* Acute upper respiratory tract infection in run-in period
* Patients who failed to achieve AR control in the run-in period
* Patients who are participating in other clinical trials
* patients who are not suitable for this clinical trial due to other reasons (evaluated by investigators).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-09-09 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
AR control level after 4-week treatment among the three groups with different treatment | 6 months
  The efficacy and safety of on-demand INS (Fluticasone) combined with nasal spray AH1(Azelastine), on-demand INS and INS maintenance therapy were evaluated and compared by recording the daily symptom score and adverse events. The primary endpoint is the AR control level after 4-week treatment.

SECONDARY OUTCOMES:
AR recurrence time after 4-week treatment | 6 months
  At the end of treatment, the patients were followed up for up to 8 weeks to compare the time interval of AR recurrence after treatment cessation (4 weeks) in the three groups.

CONTACTS AND LOCATIONS:
Overall Officials: Zheng Liu, PI, Study Director — Tongji Hospital
Locations (1):
- Tongji Hosptial affiliated to Tongji Medical college of Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes
We plan to share the periodic study reports with peers, share the data, problems we encounter in the study and problem solutions, and modification of the scheme if it is necessary.
Supporting Information: CSR
Time Frame: The Clinical Study Report (CSR) will be available in six months and for 1 year.
Access Criteria: The peer investigators who contact with the Central Contact Person by email or phone call.

REFERENCES:
- [Result] Wang XD, Zheng M, Lou HF, Wang CS, Zhang Y, Bo MY, Ge SQ, Zhang N, Zhang L, Bachert C. An increased prevalence of self-reported allergic rhinitis in major Chinese cities from 2005 to 2011. Allergy. 2016 Aug;71(8):1170-80. doi: 10.1111/all.12874. Epub 2016 Apr 13. PMID 26948849
- [Result] Claxton AJ, Cramer J, Pierce C. A systematic review of the associations between dose regimens and medication compliance. Clin Ther. 2001 Aug;23(8):1296-310. doi: 10.1016/s0149-2918(01)80109-0. PMID 11558866
- [Result] Wang Y, Zhu R, Liu G, Li W, Chen H, Daures JP, Chiriac AM, Demoly P. Prevalence of uncontrolled allergic rhinitis in Wuhan, China: a prospective cohort study. Am J Rhinol Allergy. 2014 Sep-Oct;28(5):397-403. doi: 10.2500/ajra.2014.28.4079. PMID 25198026
- [Result] Menditto E, Costa E, Midao L, Bosnic-Anticevich S, Novellino E, Bialek S, Briedis V, Mair A, Rajabian-Soderlund R, Arnavielhe S, Bedbrook A, Czarlewski W, Annesi-Maesano I, Anto JM, Devillier P, De Vries G, Keil T, Sheikh A, Orlando V, Larenas-Linnemann D, Cecchi L, De Feo G, Illario M, Stellato C, Fonseca J, Malva J, Morais-Almeida M, Pereira AM, Todo-Bom AM, Kvedariene V, Valiulis A, Bergmann KC, Klimek L, Mosges R, Pfaar O, Zuberbier T, Cardona V, Mullol J, Papadopoulos NG, Prokopakis EP, Bewick M, Ryan D, Roller-Wirnsberger RE, Tomazic PV, Cruz AA, Kuna P, Samolinski B, Fokkens WJ, Reitsma S, Bosse I, Fontaine JF, Laune D, Haahtela T, Toppila-Salmi S, Bachert C, Hellings PW, Melen E, Wickman M, Bindslev-Jensen C, Eller E, O'Hehir RE, Cingi C, Gemicioglu B, Kalayci O, Ivancevich JC, Bousquet J; MASK group. Adherence to treatment in allergic rhinitis using mobile technology. The MASK Study. Clin Exp Allergy. 2019 Apr;49(4):442-460. doi: 10.1111/cea.13333. Epub 2019 Mar 12. PMID 30597673
- [Result] May JR, Dolen WK. Management of Allergic Rhinitis: A Review for the Community Pharmacist. Clin Ther. 2017 Dec;39(12):2410-2419. doi: 10.1016/j.clinthera.2017.10.006. Epub 2017 Oct 25. PMID 29079387
- [Result] Lamb CE, Ratner PH, Johnson CE, Ambegaonkar AJ, Joshi AV, Day D, Sampson N, Eng B. Economic impact of workplace productivity losses due to allergic rhinitis compared with select medical conditions in the United States from an employer perspective. Curr Med Res Opin. 2006 Jun;22(6):1203-10. doi: 10.1185/030079906X112552. PMID 16846553
- [Result] Bedard A, Basagana X, Anto JM, Garcia-Aymerich J, Devillier P, Arnavielhe S, Bedbrook A, Onorato GL, Czarlewski W, Murray R, Almeida R, Fonseca J, Costa E, Malva J, Morais-Almeida M, Pereira AM, Todo-Bom A, Menditto E, Stellato C, Ventura MT, Cruz AA, Stelmach R, da Silva J, Larenas-Linnemann D, Fuentes-Perez JM, Huerta-Villalobos YR, Emuzyte R, Kvedariene V, Valiulis A, Kuna P, Samolinski B, Klimek L, Mosges R, Pfaar O, Shamai S, Annesi-Maesano I, Bosse I, Demoly P, Fontaine JF, Cardona V, Mullol J, Valero A, Roller-Wirnsberger RE, Tomazic PV, Chavannes NH, Fokkens WJ, Reitsma S, Bewick M, Ryan D, Sheikh A, Haahtela T, Toppila-Salmi S, Valovirta E, Makris M, Papadopoulos NG, Prokopakis EP, Psarros F, Cingi C, Gemicioglu B, Yorgancioglu A, Bosnic-Anticevich S, O'Hehir RE, Bachert C, Hellings PW, Pugin B, Bindslev-Jensen C, Eller E, Kull I, Melen E, Wickman M, De Vries G, van Eerd M, Agache I, Ansotegui IJ, Dykewicz MS, Casale T, Wallace D, Waserman S, Laune D, Bousquet J; MASK study group. Mobile technology offers novel insights into the control and treatment of allergic rhinitis: The MASK study. J Allergy Clin Immunol. 2019 Jul;144(1):135-143.e6. doi: 10.1016/j.jaci.2019.01.053. Epub 2019 Apr 3. PMID 30951790
- [Result] Bateman ED, Reddel HK, O'Byrne PM, Barnes PJ, Zhong N, Keen C, Jorup C, Lamarca R, Siwek-Posluszna A, FitzGerald JM. As-Needed Budesonide-Formoterol versus Maintenance Budesonide in Mild Asthma. N Engl J Med. 2018 May 17;378(20):1877-1887. doi: 10.1056/NEJMoa1715275. PMID 29768147
- [Result] O'Byrne PM, FitzGerald JM, Bateman ED, Barnes PJ, Zhong N, Keen C, Jorup C, Lamarca R, Ivanov S, Reddel HK. Inhaled Combined Budesonide-Formoterol as Needed in Mild Asthma. N Engl J Med. 2018 May 17;378(20):1865-1876. doi: 10.1056/NEJMoa1715274. PMID 29768149
- [Result] Bousquet J, Khaltaev N, Cruz AA, Denburg J, Fokkens WJ, Togias A, Zuberbier T, Baena-Cagnani CE, Canonica GW, van Weel C, Agache I, Ait-Khaled N, Bachert C, Blaiss MS, Bonini S, Boulet LP, Bousquet PJ, Camargos P, Carlsen KH, Chen Y, Custovic A, Dahl R, Demoly P, Douagui H, Durham SR, van Wijk RG, Kalayci O, Kaliner MA, Kim YY, Kowalski ML, Kuna P, Le LT, Lemiere C, Li J, Lockey RF, Mavale-Manuel S, Meltzer EO, Mohammad Y, Mullol J, Naclerio R, O'Hehir RE, Ohta K, Ouedraogo S, Palkonen S, Papadopoulos N, Passalacqua G, Pawankar R, Popov TA, Rabe KF, Rosado-Pinto J, Scadding GK, Simons FE, Toskala E, Valovirta E, van Cauwenberge P, Wang DY, Wickman M, Yawn BP, Yorgancioglu A, Yusuf OM, Zar H, Annesi-Maesano I, Bateman ED, Ben Kheder A, Boakye DA, Bouchard J, Burney P, Busse WW, Chan-Yeung M, Chavannes NH, Chuchalin A, Dolen WK, Emuzyte R, Grouse L, Humbert M, Jackson C, Johnston SL, Keith PK, Kemp JP, Klossek JM, Larenas-Linnemann D, Lipworth B, Malo JL, Marshall GD, Naspitz C, Nekam K, Niggemann B, Nizankowska-Mogilnicka E, Okamoto Y, Orru MP, Potter P, Price D, Stoloff SW, Vandenplas O, Viegi G, Williams D; World Health Organization; GA(2)LEN; AllerGen. Allergic Rhinitis and its Impact on Asthma (ARIA) 2008 update (in collaboration with the World Health Organization, GA(2)LEN and AllerGen). Allergy. 2008 Apr;63 Suppl 86:8-160. doi: 10.1111/j.1398-9995.2007.01620.x. No abstract available. PMID 18331513
- [Result] Wang J, Wu Y, Li J, Huang X, Zhu R. Eight Aeroallergen Skin Extracts May Be the Optimal Panel for Allergic Rhinitis Patients in Central China. Int Arch Allergy Immunol. 2017;173(4):193-198. doi: 10.1159/000479429. Epub 2017 Aug 29. PMID 28848100
- [Result] Demoly P, Jankowski R, Chassany O, Bessah Y, Allaert FA. Validation of a self-questionnaire for assessing the control of allergic rhinitis. Clin Exp Allergy. 2011 Jun;41(6):860-8. doi: 10.1111/j.1365-2222.2011.03734.x. Epub 2011 Apr 25. PMID 21518040
- [Result] Zhu R, Wang J, Wu Y, Yang Y, Huang N, Yang Y, Zhang R, Ma D, Yang L, Demoly P. The Allergic Rhinitis Control Test Questionnaire Is Valuable in Guiding Step-Down Pharmacotherapy Treatment of Allergic Rhinitis. J Allergy Clin Immunol Pract. 2019 Jan;7(1):272-278. doi: 10.1016/j.jaip.2018.05.028. Epub 2018 Jun 7. PMID 29886146
- [Result] Wang Y, Chen H, Zhu R, Liu G, Huang N, Li W, Yang L, Zhang S, Qi S, Daures JP, Chiriac AM, Demoly P. Allergic Rhinitis Control Test questionnaire-driven stepwise strategy to improve allergic rhinitis control: a prospective study. Allergy. 2016 Nov;71(11):1612-1619. doi: 10.1111/all.12963. Epub 2016 Jul 20. PMID 27332957
- [Result] Bachert C, Bousquet J, Hellings P. Rapid onset of action and reduced nasal hyperreactivity: new targets in allergic rhinitis management. Clin Transl Allergy. 2018 Jun 25;8:25. doi: 10.1186/s13601-018-0210-2. eCollection 2018. PMID 29983907
- [Result] Wartna JB, Bohnen AM, Elshout G, Pijnenburg MW, Pols DH, Gerth van Wijk RR, Bindels PJ. Symptomatic treatment of pollen-related allergic rhinoconjunctivitis in children: randomized controlled trial. Allergy. 2017 Apr;72(4):636-644. doi: 10.1111/all.13056. Epub 2016 Oct 28. PMID 27696447
- [Result] Zheng YW, Lai XX, Zhao DY, Zhang CQ, Chen JJ, Zhang L, Wei QY, Chen S, Liu EM, Norback D, Gjesing B, Zhong NS, Spangfort DM. Indoor Allergen Levels and Household Distributions in Nine Cities Across China. Biomed Environ Sci. 2015 Oct;28(10):709-17. doi: 10.3967/bes2015.101. PMID 26582093